CLINICAL TRIAL: NCT02044744
Title: Primary Care Physical Activity Referrals to the Community
Brief Title: Physical Activity Referrals to the Community
Acronym: PARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-08-5557; 035156 (Other Grant/Funding Number: Safeway Foundation)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Overweight; Obesity
Keywords: Obesity; Pediatric Obesity; Physical Activity; Physical Fitness; Primary Health Care; Referral and Consultation
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Referral (Experimental): Physical activity referral
  Interventions: Behavioral: Physical activity referral
- Wait-list control (No Intervention): Wait-list controls receive no intervention until after they provide follow-up measurements.

INTERVENTIONS:
Behavioral: Physical activity referral — Provision of a primary care referral to at least one community-based physical activity program that is a good match for the participant's needs and preferences and patient follow-up on enrollment.
  Arms: Referral

SUMMARY:
The purpose of this study is to determine the impact of primary care referrals to community physical activity programs for overweight and obese youth aged 6-18 years on objectively measured physical activity and cardiorespiratory fitness, as well as other cardiovascular health indicators. We hypothesize that physical activity referrals will result in higher levels of physical activity and fitness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-18 years
* Body mass index greater than or equal to the 85th percentile for age and sex or greater than or equal to 25 for youth aged 18
* Fluent in English
* Parent of participant must be fluent in either English or Spanish

Exclusion Criteria:

* Medical conditions that preclude participation in physical activity

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in minutes per day of moderate-to-vigorous physical activity | Baseline and at 8-11 weeks
  Assessed via accelerometry
Change in cardiorespiratory fitness | Baseline and at 10-12 weeks
  Assessed via 3 minute step test

SECONDARY OUTCOMES:
Change in body mass index | Baseline and at 10-12 weeks
Change in body composition | Baseline and at 10-12 weeks
Change in blood pressure | Baseline and at 10-12 weeks

OTHER OUTCOMES:
Enrollment and participation in a physical activity program | Baseline and at 10-12 weeks
Change in waist circumference | Baseline and at 10-12 weeks
Change in perceptions about physical activity | Baseline and at 10-12 weeks
  Assessed via survey

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Madsen, MD, MPH, Principal Investigator — University of California, Berkeley
Locations (4):
- United States (4):
  - Healthy Lifestyles, San Francisco General Hospital, San Francisco, California
  - Mission Neighborhood Health Center, San Francisco, California
  - Southeast Health Center, San Francisco, California
  - Silver Avenue Health Center, San Francisco, California